CLINICAL TRIAL: NCT01887561
Title: PhaseⅡClinical Trial of Dasatinib for Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase and Stop Therapy After Achieving Complete Molecular Response for Cure D-NewS
Brief Title: Dasatinib for Patients Achieving Complete Molecular Response for Cure D-NewS Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanto CML Study Group (Other)
Responsible Party: Principal Investigator, Naoki Takezako, M.D., Ph.D., Kanto CML Study Group, Kanto CML Study Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-04
Record Dates: First submitted 2013-04-11; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Myelogenous Leukemia, Chronic, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (No Intervention)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib

SUMMARY:
The purpose of this study is to assess whether dasatinib can be discontinued without occurrence of molecular relapse in patients with chronic myeloid leukemia in chronic phase in complete molecular remission(CMR) while on dasatinib.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Chronic Myeloid Leukemia in the Chronic Phase
* 15 years old over.
* ECOG performance status (PS) score 0-2.
* Adequate organ function (hepatic, renal and lung).
* Signed written informed consent.

Exclusion Criteria:

* A case with the double cancer of the activity.
* Women who are pregnant or breastfeeding.
* female patient who there is not intention with an appropriate sterilization, or cannot use it during a study entry period
* Patients with complications or a history of severe or uncontrolled cardiovascular failure following have a Myocardial infarction within 6 months have an Angina within 3 months have a Congestive heart failure within 3 months have a QTc interval of more than 450msec at baseline
* A serious uncontrolled medical disorder that would impair the ability of the subjects to receive protocol therapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The overall probability of maintenance of complete molecular remission after stopping dasatinib as measured by RQ-PCR | by 12 months

SECONDARY OUTCOMES:
'Dasatinib affects immunological responses, as measured by flow cytometry | at 3,6,12,24 months
Major Molecular Response(MMR) rate measured by RQ-PCR | by 1 months, then every 6 months for 2 years
Complete Cytogenetic Response (CCyR) rate | by 6,12 months
Progression free survival (PFS) | Participants were followed for at least 2 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Participants were followed for at least 2 years
The overall probability of maintenance of complete molecular remission after stopping dasatinib as measured by RQ-PCR | by 3,6 months
Molecular remission rate measured by PQ-PCR after dasatinib re-challenge in cases of molecular relapse | by 12 months after molecular relapse
Complete Molecular Response(CMR) rate measured by RQ-PCR | by 1 months, then every 6 months for 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Disaster Medical Center, Tachikawa, Tokyo, Japan